CLINICAL TRIAL: NCT02862028
Title: A Clinical Study of PD-1 Antibody Expressing CAR-T Cells for EGFR Family Member Positive Advanced Solid Tumor (Lung, Liver and Stomach)
Brief Title: PD-1 Antibody Expressing CAR-T Cells for EGFR Family Member Positive Advanced Solid Tumor (Lung, Liver and Stomach)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai International Medical Center (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIMC-20160101/02/03
Record Dates: First submitted 2016-08-07; First posted 2016-08-10 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: PD-1 Antibody; CAR-T Cells; Advanced Solid Tumor
Keywords: PD-1 antibody; CAR-T cells; EGFR family; advanced solid tumor

ARMS (1):
- HerinCAR-PD1 cells (Experimental): Patients will receive 3 cycles of HerinCAR-PD1 cells treatment.
  Interventions: Biological: HerinCAR-PD1 cells

INTERVENTIONS:
Biological: HerinCAR-PD1 cells — herinCAR-PD1 cells transfusion: (1-5×107/kg herinCAR-PD1 + physiological saline + 0.25% human alloalbumin) 300ml for each infusion. IV (in the vein) for each infusion, 2 cycles, each cycle received one infusions on day 21, 43.

SUMMARY:
Objectives:

To evaluate the safety and effectiveness of cell therapy using herinCAR-PD1 cells to treat relapsed or refractory cancer.

Eligibility:

Individuals greater than or equal to 18 years of age and less than or equal to 70 years of age who have been diagnosed with relapsed or refractory cancer that has not responded to or has relapsed after standard treatment.

DETAILED DESCRIPTION:
A total of 20 patients may be enrolled over a period of 1-2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18~65 years old, male or female;
2. Life expectancy≥6 months;
3. ECOG score: 0-3;
4. Advanced solid tumor (lung cancer, gastric cancer, liver cancer) were diagnosed by pathological or clinical physicians;
5. Enough venous channel, no other contraindications to the separation and collection of white blood cells;
6. Immunohistochemistry and RT-PCR technology will be used to determine the positive EGFR family (including EGFR, HER2, HER4) and IGFR1 protein. At least one protein expressed in immunohistochemical tumor tissue should be no less than grade 2 or 2+ scores. The levels of protein are defined as follows: (according to cell staining) : grade 0: without staining; grade 1: 1-25%; grade 2: 26-50% and grade 3: 51-100%; (According to the intensity): negative; 1+; 2+ and 3+;
7. Laboratory examination: white blood cell≥3 x 10*9/L, blood platelet count≥60 x 10*/L, hemoglobin≥85g/L; lymphocyte count≥15%, total bilirubin≤100 mol/L; ALT and AST less than five times of the normal level; serum creatinine less than 1.5 times of the normal level；
8. Signed informed consent；
9. Women of child-bearing age must have evidence of negative pregnancy test and be willing to practice birth control after 2 weeks following the cells transfusion.

Exclusion Criteria:

1. Expected Overall survival < 6 months;
2. Patients with uncontrolled hypertension, unstable coronary disease (uncontrolled arrhythmias, unstable angina, decompensated congestive heart failure (> Class II, NYHA), or myocardial infarction within 6 months.
3. Abnormal lung function: FEV (forced expiratory volume) < 30% prediction, DLCO (diffusing capacity of the lung for carbon monoxide) < 30% prediction, blood oxygen saturation < 90%;
4. Other serious diseases: nervous, mental disorders, immune regulatory diseases, metabolic diseases, infectious diseases, etc;
5. Unable or unwilling to provide informed consent, or fail to comply with the test requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-03 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 2 years
Disease control rate,(DCR) | 2 years
Overall survival | 2 years
Progress-free survival(PFS) | 2 years

SECONDARY OUTCOMES:
Quality of life | 2 years
  Questionnaire will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Naiyan Han, Study Chair — Shanghai International Medical Center
Locations (1):
- Shanghai International Medical Center, Shanghai, Shanghai Municipality, China